CLINICAL TRIAL: NCT05514561
Title: Diagnostic Performance of Fecal Immunochemical Test and Fecal Calprotectin in Detection of Ileocolonic Lesions in Patients With Chronic Lower Gastrointestinal Symptoms
Brief Title: FIT and Fecal Calprotectin in Patients With Chronic Lower GI Symptoms
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Julajak Limsrivilai, Associate Professor, Mahidol University
Other Study IDs: Si238/2020
Record Dates: First submitted 2022-05-24; First posted 2022-08-24 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Colorectal Cancer; Colorectal Adenoma; Colitis
Keywords: Fecal immunochemical test; calprotectin; Colorectal neoplasm; Colorectal cancer; Colitis
MeSH Terms: conditions — Colorectal Neoplasms; Colitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with chronic lower gastrointestinal symptoms: We enroll adults older than 18 years with chronic lower GI symptoms for more than 1 month and are scheduled for a colonoscopy. The lower GI symptoms consist of any of the followings; lower abdominal pain, constipation, diarrhea, rectal bleeding, change in stool caliber, and abdominal bloating.
  Interventions: Diagnostic Test: Fecal calprotectin; Diagnostic Test: Fecal immunochemical test

INTERVENTIONS:
Diagnostic Test: Fecal calprotectin — To calculate the diagnostic accuracy of fecal calprotectin in the diagnosis of significant ileocolonic lesions
Diagnostic Test: Fecal immunochemical test — To calculate the diagnostic accuracy of the fecal immunochemical test in the diagnosis of significant ileocolonic lesions

SUMMARY:
Chronic lower gastrointestinal (GI) symptoms, including lower abdominal pain, bowel habit change, bleeding per rectum, and abdominal bloating, are caused by functional gastrointestinal disorders (FGID) and organic intestinal disorders, including colorectal cancer and chronic colitis. The presence of alarming features, such as the age of onset older than 50 years, rectal bleeding, anemia, significant weight loss, and family history of colorectal cancer, indicates organic diseases, and colonoscopy should be required. However, using only alarming features may not be sufficiently accurate. For example, anemia or significant weight loss, which are highly specific for organic disorders, usually occur in late-stage diseases. Conversely, the parameters with high sensitivity, such as the age of onset after 50 years, have a low specificity; colonoscopy in these patients may not be urgent. Therefore, tests that can help discriminate organic from functional diseases are warranted. Immunochemical fecal occult blood tests (iFOBT) and fecal calprotectin (FC) are biomarkers that indicate organic lesions in the gastrointestinal tract and could help diagnose patients with lower GI symptoms more accurately.

DETAILED DESCRIPTION:
This study was a single-center, prospective cohort study undertaken at Siriraj hospital between March 2020 to November 2022. Eligible participants were required to collect their stool samples one to two days before the bowel preparation. The stool was sent for fresh smear examination, quantitative FIT (OC-SENSOR, EIKEN CHEMICAL, Japan), and quantitative fecal calprotectin (EliA Calprotectin 2, Phadia, Sweden). Blood samples were obtained on the day of the colonoscopy and were tested for complete blood count, albumin, and C-reactive protein (CRP) levels. In addition, clinical information was obtained, including alarm features such as the age of onset older than 50 years, rectal bleeding, anemia, significant weight loss, and family history of colorectal cancer. Colonoscopic findings and histopathological findings were used as the reference standard for diagnosis. We analyzed the sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) for diagnosing significant ileocolonic lesions, including colorectal cancer, advanced adenoma, and colitis, of each diagnostic modality comparing to the reference standard.

ELIGIBILITY:
Inclusion criteria

* age of at least 18 years
* patients with at least one month of any lower gastrointestinal symptoms are as followings; lower abdominal pain, constipation, diarrhea, rectal bleeding, change in stool caliber, abdominal bloating,
* patients who are scheduled for a colonoscopy

Exclusion criteria

* incomplete colonoscopy
* incomplete stool collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We enrolled adults older than 18 years with chronic lower GI symptoms for more than 1 month and were scheduled for a colonoscopy. The lower GI symptoms consisted of any of the followings; lower abdominal pain, constipation, diarrhea, rectal bleeding, change in stool caliber, and abdominal bloating. The stool samples were collected one to two days before the bowel preparation. All patients provided written informed consent. Patients who did not return their stool samples and whose complete colonoscopy was not achieved were excluded.
Sampling Method: Probability Sample
Enrollment: 1007 (Actual)
Dates: Start 2020-03-22 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
The diagnostic performance of fecal calprotectin in diagnosis of significant ileocolonic lesions | 1 month
  The sensitivity, specificity, and accuracy of fecal calprotectin in diagnosis of significant ileocolonic lesions, including colorectal cancer, advanced adenoma, and ileocolitis, compared to colonoscopic diagnosis

SECONDARY OUTCOMES:
The diagnostic performance of fecal immunochemical test in diagnosis of significant ileocolonic lesions | 1 month
  The sensitivity, specificity, and accuracy of fecal immunochemical test in diagnosis of significant ileocolonic lesions, including colorectal cancer, advanced adenoma, and ileocolitis, compared to colonoscopic diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Julajak Limsrivilai, MD, MS, Principal Investigator — Siriraj Hospital
Locations (1):
- Gastroenterology division, Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Limsrivilai J, Yodmalai C, Chaemsupaphan T, Sattayalertyanyong O, Subdee N, Permpim P, Phaophu P, Kaosombatwattana U, Pausawasdi N, Riansuwan W, Charatcharoenwitthaya P, Pongprasobchai S. Evaluating the Efficacy of Fecal Immunochemical Test, Fecal Calprotectin, and Serum C-Reactive Protein in Diagnosing Patients With Chronic Lower Gastrointestinal Symptoms. Clin Transl Gastroenterol. 2024 Aug 1;15(8):e00747. doi: 10.14309/ctg.0000000000000747. PMID 38994833